CLINICAL TRIAL: NCT06571721
Title: Prospective, Double-Blinded, Randomized Study of Topical Almond Oil and Tretinoin on Facial Wrinkles
Brief Title: The Effects of Topical Almond Oil and Tretinoin on Facial Wrinkles
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Integrative Skin Science and Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRI24_01_AlmondOil
Record Dates: First submitted 2024-08-23; First posted 2024-08-26 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Collagen Degeneration; Wrinkle; Pigmentation; Elastic Skin; Sebum Deficiency
Keywords: Facial Wrinkles; Skin biophysical properties; Photoaging; Pigmentation
MeSH Terms: conditions — Ehlers-Danlos Syndrome | interventions — Vitamin E; Pharmaceutical Preparations; Castor Oil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Almond Oil (Experimental): Almond Oil. 1-2 Drops of randomized topical product will be applied on entire face nightly. Duration: 16 weeks
  Interventions: Other: Topical Product: Almond Oil
- Almond oil augmented with 0.5% Vitamin E (Experimental): Almond oil augmented with 0.5% Vitamin E. 1-2 Drops of randomized topical product will be applied on entire face nightly. Duration: 16 weeks
  Interventions: Other: Topical Product: Almond oil augmented with 0.5% Vitamin E
- 0.025% Tretinoin oil augmented with castor oil (Experimental): 0.025% Tretinoin oil augmented with castor oil. 1-2 Drops of randomized topical product will be applied on entire face nightly. Duration: 16 weeks
  Interventions: Other: Topical Product: 0.025% Tretinoin oil augmented with castor oil

INTERVENTIONS:
Other: Topical Product: Almond Oil — 1-2 Drops of randomized topical product will be applied on entire face nightly.
  Arms: Almond Oil
Other: Topical Product: Almond oil augmented with 0.5% Vitamin E — 1-2 Drops of randomized topical product will be applied on entire face nightly.
  Arms: Almond oil augmented with 0.5% Vitamin E
Other: Topical Product: 0.025% Tretinoin oil augmented with castor oil — 1-2 Drops of randomized topical product will be applied on entire face nightly.
  Arms: 0.025% Tretinoin oil augmented with castor oil

SUMMARY:
Investigate the topical use of almond oil, almond oil augmented with 0.5% vitamin E, 0.025% tretinoin oil augmented with castor oil on the appearance of facial fine lines and wrinkles, pigmentation, hydration, trans-epidermal water loss, and sebum excretion rate.

DETAILED DESCRIPTION:
The natural cosmetic market is a multi-billion dollar industry. Nutraceuticals and food-based cosmetics are a growing trend within dermatology. Almonds are a rich dietary source of a range of fatty acids, phytochemical polyphenols, and antioxidants. Our previous study was a double blinded study that compared almond consumption interventions to a calorie matched intervention over 16 weeks. The study determined that that there was a statistically significant 8.41% improvement in wrinkle severity in the women that received almond supplementation. This proposal aims to now understand how the topical application of almond oil may influence the appearance of wrinkles and facial tone in post-menopausal women. Almond oil is rich in fatty acids and alpha-tocopherol. Tocopherol inhibits melanogenesis in melanocytes and topical alpha tocopherol has been shown to improve skin antioxidants and hyperpigmentation. A challenge of almond oil is that it is prone to oxidation due to its high unsaturated fatty acid concentrations. However, tocopherol has also been shown to improve almond oil stability.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women of Fitzpatrick skin types 1, 2, and 3
* Individuals with facial fine lines and wrinkles

Exclusion Criteria:

* Individuals who are pregnant or breastfeeding
* Prisoners
* Adults unable to consent
* Those with a nut allergy or tocopherol allergy
* Current smokers, those that have smoked within the past year, and former smokers with greater than a 10-pack- year history of smoking
* Those with an autoimmune photosensitive condition or a known genetic condition with a deficiency in collagen production (such as Ehlers-Danlos syndromes)
* Those who have undergone any cosmetic procedures to the face in the 3 months prior to enrollment in the opinion of the investigator. People that have undergone deeper chemical peels (TCA based peels) within 1 year prior to enrollment
* Individuals who are unwilling to discontinue vitamin E containing supplements and food sources such as all nuts, sunflower seeds or sunflower oil during the washout and intervention
* Individual who are unwilling to discontinue topical cosmetic products during the duration of the study or unwilling to undergo a 2-week washout of topicals that are known to modulate collagen and pigment:
* Retinoids such as tretinoin, adapalene, retinol, except as provided by the study.
* Antioxidant ingredients such as vitamin C or vitamin E.
* Pigment reducing agents such as hydroquinone, azelaic acid, kojic acid, or a retinoid except for the retinol that is provided in this study.
* Topicals that contain a nut oil or nut extract as part of their ingredient list.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-01-22 (Estimated); Study Completion 2025-07-22 (Estimated)

PRIMARY OUTCOMES:
Facial wrinkles | 16 Weeks
  Change in severity of wrinkles measured by photographic analysis (BTBP 3D Camera System)

SECONDARY OUTCOMES:
Changes in Pigment intensity through the use of high resolution photography (BTBP Clarity Pro) | 16 Weeks
  Change in the appearance of facial pigmentation by high resolution photography (BTBP Clarity Pro) and measures intensity of facial pigmentation. Higher scores indicate darker pigmentation.
Pigment intensity measured through SkinColorCatch. | 16 Weeks
  Change in the appearance of facial pigmentation will be measured on both cheeks through the use of a handheld device known as the SkinColorCatch with quantitative output for pigment intensity.
Changes in skin hydration | 16 Weeks
  Change in skin hydration will be measured on both cheeks through the use of a non-invasive device known as the Moisturemeter.
Sebum excretion rate | 16 Weeks
  Measure of skin sebum via sebumeter
Tolerability Assessment Questionnaire | 16 Weeks
  A 6 question survey based on the self-assessment about the tolerability of the topical skin product. The scale ranges from 0-3 with 0 being the best outcome possible and with 3 being the worst. "0" as none, "1" as mild, "2" as moderate, or "3" as severe.
Transepidermal water loss | 16 Weeks
  Change in transepidermal water loss (TEWL) using the Vapometer

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Research Institute, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No